CLINICAL TRIAL: NCT05839379
Title: Molecularly-Guided Phase II Umbrella Trial for Children, Adolescents, and Young Adults Newly Diagnosed With High-Grade Glioma, Including Diffuse Intrinsic Pontine Glioma
Brief Title: Targeted Pediatric High-Grade Glioma Therapy
Status: Recruiting | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CONNECT TarGeT-SCR; R01FD008167 (FDA)
Record Dates: First submitted 2023-04-20; First posted 2023-05-03 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-09

CONDITIONS: High Grade Glioma; Diffuse Intrinsic Pontine Glioma; Anaplastic Astrocytoma; Glioblastoma; Glioblastoma Multiforme; Diffuse Midline Glioma, H3 K27M-Mutant; Metastatic Brain Tumor; WHO Grade III Glioma; WHO Grade IV Glioma
MeSH Terms: conditions — Glioma; Diffuse Intrinsic Pontine Glioma; Astrocytoma; Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Brain tumor samples with matched normal comparator (blood preferred alternatively, saliva or buccal swab)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to perform genetic sequencing on brain tumors from children, adolescents, and young adult patients who have been newly diagnosed with a high-grade glioma. This molecular profiling will decide if patients are eligible to participate in a subsequent treatment-based clinical trial based on the genetic alterations identified in their tumor.

DETAILED DESCRIPTION:
A novel, molecularly-guided, multi-arm phase umbrella II trial is proposed in children, adolescents, and young adults with newly diagnosed HGG, including DIPG, in which we will (1) conduct comprehensive molecular screening of tumor tissue using a multi-omic approach (WES/WGS, gene fusion panels/RNASeq, DNA methylation microarray) across international CONNECT genomics cores with rapid return of clinical results, (2) stratify patients to biologically-targeted treatment arms, based on the tumor molecular profile and histopathology, and (3) perform longitudinal evaluation of peripheral blood, cerebrospinal fluid (CSF), and/or tumor tissue as well as advanced neuro-imaging to determine genomic, immune, and radiologic biomarkers predictive of response, recurrence, resistance, and toxicity.

Based on results of the above tumor molecular profiling and pathology-based confirmation of HGG diagnosis, eligible patients will be assigned to one of several biologically guided treatment arms on a phase II trial.

Approximately 300-350 patients will be enrolled on the screening protocol through which biospecimens (paired tumor DNA/RNA and normal comparator samples) will undergo extensive molecular profiling and/or there will be comprehensive central molecular and pathology review of previously obtained molecular results to assess eligibility to any of the therapeutic subprotocols of the phase II study.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Patients must be ≥12 months and ≤39 years of age at the time of enrollment onto this screening protocol.
2. Diagnosis: Patients with newly diagnosed HGG, including DIPG are eligible. Diagnosis must have histologic confirmation from biopsy or resection. The diagnosis of HGG must have been confirmed by pathology review at the local site. For the diagnosis of DIPG, patients must have a tumor with pontine epicenter and diffuse involvement of at least 2/3 of the pons, with histopathology consistent with diffuse WHO grade 2-4 glioma (eg, diffuse astrocytoma, anaplastic astrocytoma, glioblastoma, H3K27-altered diffuse midline glioma). For all other tumors, histologic grade must be WHO grade 3-4.
3. Disease Status: There are no disease status requirements for enrollment.

   * Measurable disease is not required. Patients without measurable disease are eligible.
   * Patients with metastatic/disseminated or multifocal disease or gliomatosis cerebri are eligible.
   * Patients with a primary spinal tumor are eligible.
   * Patients with secondary, radiation related HGG are eligible.
4. Prior Therapy for HGG: Surgery, radiation, and/or dexamethasone are permissible. Temozolomide concurrent with radiation is permissible. Prior administration of avastin/bevacizumab is allowed (individual treatment arms have different washout period requirements, check individual arm eligibility). No other prior anticancer therapy for HGG will be allowed.

   * Participants screening for assignment to TarGeT-L may not have received radiation.

   Timing from surgery to start of RT: For patients who have started RT, radiation must have started <42 days from definitive surgery or biopsy, however it is strongly recommended patients start RT within 31 days from definitive surgery (if patient had two surgeries, radiation must have started within 31 days from second surgery).
5. Tumor Sample Availability OR results from previous molecular profiling/targeted sequencing

   * If a patient screens through OPTION #1, tumor sample in addition to normal comparator tissue (peripheral blood, saliva, or buccal swab) must be submitted for comprehensive molecular screening at the time of screening enrollment.
   * If a patient screens through OPTIONS #2 or #3, results from previously performed molecular profiling must be submitted following enrollment. It is highly recommended that results be uploaded within 7 days of enrollment (if results are available at time of enrollment) or within 7 days of results becoming available (if pending at time of enrollment) to allow adequate time for central review.
6. Informed Consent: All patients and/or their parents or legally authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.
7. Enrollment timeline: Patients are eligible to enroll on the TarGeT-SCR anytime between diagnosis and the following specific timepoints post completion of RT (if relevant)

   * Patients screening through OPTION #1 are eligible to enroll anytime between diagnosis and 10 days post RT (if completing RT).
   * Patients screening through OPTIONS #2 or #3 are eligible to enroll anytime between diagnosis and 21 days post RT (if completing RT).
   * Participants screening for TarGeT-L (lorlatinib) are eligible to enroll on TarGeT-SCR anytime between diagnosis and 31 days post definitive surgery (to allow time for molecular review).

However, it is important to note the following:

* For treatment protocols that include targeted therapy administered concurrently with RT, patients must start treatment within 10 calendar days of starting RT.
* For treatment protocols that only include maintenance/adjuvant therapy (no systemic therapy given concurrently with radiation), patients must start treatment by 35 days post RT

  #SCREENING OPTIONS
* OPTION1: Molecular screening through CONNECT TarGeT Clinical Testing Laboratories
* OPTION2: Molecular screening through a national comprehensive tumor profiling program
* OPTION3: Clinically validated targeted sequencing or focused profiling

Exclusion Criteria:

-Tumors that do not meet HGG and DIPG diagnoses specified above

Ages: 12 Months to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric and young adult patients new diagnosed with High Grade Glioma including Diffuse Intrinsic Pontine Glioma (per 2021 WHO CNS tumor classification)
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2029-08-28 (Estimated); Study Completion 2034-08-28 (Estimated)

PRIMARY OUTCOMES:
Molecular profiling | 4 years
  Utilize molecular, clinical, and histopathologic data to assess eligibility for specific biologically-guided treatment subprotocols among pediatric, adolescent and young adult patients with newly diagnosed HGG, including DIPG.
Feasibility of molecular profiling and enrollment to a TarGeT treatment protocol | 4 years
  Determine the percent of pediatric, adolescent, and young adult patients newly diagnosed with HGG, including DIPG, who undergo screening through one of three TarGeT-SCR screening mechanisms and are assigned to a TarGeT treatment arm.

SECONDARY OUTCOMES:
Genomic Research | 6 years
  Increase knowledge of the genomic and immunologic landscape of newly-diagnosed pediatric and young adult HGGs, including DIPG, through comprehensive molecular characterization.
Germline susceptibility testing | 4 years
  Determine the frequency and spectrum of germline cancer susceptibility mutations in children and young adults with HGG and DIPG and assess the feasibility of return of those results.
Biobanking | 4 years
  Prospectively collect tumor tissue from diagnostic biopsy/resection as well as baseline peripheral blood and cerebrospinal fluid (CSF) samples for the CONNECT biorepository to be used in correlative research for the present trial as well as future studies.
Progression Free Survival | 4 years
  Prospectively collect data to estimate the distribution of PFS in HGG and DIPG patients, respectively, who do not enroll on any TarGeT treatment subprotocol.
Feasibility of Assignment | 4 years
  Determine the percent of pediatric, adolescent, and young adult patients newly diagnosed with HGG, including DIPG, who are assigned to a TarGeT treatment arm through one of the three TarGeT-SCR screening mechanisms, and begin treatment on a TarGeT treatment subprotocol within the required timelines.
Descriptively analyze patients not assigned | 4 years
  For patients who consent to TarGeT-SCR but do not enroll on a TarGeT treatment subprotocol: Descriptively capture and analyze reasons for lack of treatment arm enrollment.
Overall Survival | 4 years
  Prospectively collect data to estimate the distribution of OS in HGG and DIPG patients, respectively, who do not enroll on any TarGeT treatment subprotocol.

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Fouladi, MD, Study Chair — Nationwide Children's Hospital; Margot Lazow, MD, Study Director — Nationwide Children's Hospital
Locations (21):
- United States (11):
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Duke University Health System, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Australia (4):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Royal Children's Hospital, Melbourne, Victoria
  - Perth Children's Hospital, Perth, Western Australia
- Canada (2):
  - The Hospital for Sick Children (SickKids), Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
- Hopp Children's Cancer Center at NCT Heidelberg (KiTZ), Heidelberg, Baden-Wurttemberg, Germany
- Princess Máxima Center, Utrecht, Netherlands
- Starship Children's Hospital, Auckland, Grafton, New Zealand
- Great Ormond Street Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided